CLINICAL TRIAL: NCT06803771
Title: A Randomised Trial to Evaluate the cfDNA Pancreatic Cancer Test (Avantect) in the Early Detection of Pancreatic Cancer in Patients With Newly Diagnosed Diabetes Mellitus
Brief Title: Surveillance of Pancreatic Health After Diabetes Diagnosis
Acronym: SAFE-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: ClearNote Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RHMGSU0292
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus; Pancreatic Cancer, Adult
Keywords: Type 2 diabetes; pancreatic cancer
MeSH Terms: conditions — Diabetes Mellitus; Pancreatic cancer, adult; Diabetes Mellitus, Type 2; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be blindly randomised in 1:1 ratio to either the intervention arm or the control arm.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention Arm will have their blood samples tested on the Avantect test within prioritised timeframe. The "detected" Avantect test results will be shared with the participants and their General Practitioners (GPs) to allow for further MRI or CT investigations by the local clinical team.
  Interventions: Device: Avantect Pancreatic Cancer Test
- Control Arm (Standard of Care [SoC] arm) (Placebo Comparator): Control arm participants will have their blood samples collected but they will not be tested on the Avantect test. Participants will receive the current standard of care for diabetes management. Blood samples will be used for potential future Avantect testing and/ or future research.
  Interventions: Device: Avantect Pancreatic Cancer Test

INTERVENTIONS:
Device: Avantect Pancreatic Cancer Test — Avantect test

SUMMARY:
The goal of this interventional study is to evaluate if the novel diagnostic blood test, called Avantect can early detect pancreatic cancer in patients diagnosed with type 2 diabetes within the last 6 months.

Participants will:

* attend 3 study visits over 12 months time
* provide a blood sample at each study visit
* complete an anxiety questionnaire at each visit.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is one of the most lethal common cancers (five-year survival 5-7%). In more than 80% of patients the disease has spread before it is detected, ruling out potentially curative treatment options. Early detection offers the possibility of surgery leading to significantly improved overall survival.

There is currently no accepted screening test for pancreatic cancer. The Aventect test is designed to detect clues, or biomarkers for the presence or absence of pancreatic cancer signals in blood. The SAFE-D study will evaluate if the Avantect test can detect pancreatic cancer at an earlier more treatable stage.

People older than 50 years who have recently been diagnosed with type II diabetes have up to ten times higher-than-average risk of having pancreatic cancer without knowing.

The study will recruit up to 15,000 participants aged 50-84 years old diagnosed with type II diabetes within the last 6 months from GP practices over 3 years.

Participants will be randomly assigned to either the active intervention arm or the control arm for comparison. Intervention arm samples will be run on the Avantect test as soon as possible. If a pancreatic biomarker is detected the participants will be informed and offered a standard of care diagnostic imaging scan (MRI or CT) to rule out pancreatic cancer. Control arm samples will be stored for potential future Avantect testing or future research. All participants will be followed remotely via cancer and mortality registry searches for 3 years from consent to assess any cancer diagnosed during this time.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 84 years of age at the time of enrolment (within year of birth, not month of birth)
* Haemoglobin A1c (HbA1c) ≥ 48 or 6.5% and/or confirmed type II DM diagnosed within the last 180 days (+20 days flexibility allowance)
* Willing to provide up to 30 mL of blood for each study visit
* Willing and eligible to undergo MRI scan (or CT scan if MRI is contraindicated)
* Understands the study process and is willing to take part in the study and sign the informed consent form

Exclusion Criteria:

* Prior type I or type II DM diagnosis > 6 months
* A history of pancreatic cancer, pancreatic neuroendocrine tumour (pNET) or Pancreatitis
* Under investigation for pancreatic cancer / pancreatic cyst
* Any known pancreatic surgery (not including ERCP), or other major surgery requiring anaesthesia within 3 months
* Any invasive solid or haematological cancer in the past 3 years, including cancer recurrence after treatment in the last 3 years
* Current chronic or acute oral or systemic steroid use within 3 months of initial HbA1c or diabetes diagnosis (estimate rather than accurate)
* Blood transfusion within 1 month
* Solid organ transplant recipient
* Currently pregnant
* Needing dialysis

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Avantect test | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  The proportion of participants in the intervention arm with one (or more) Avantect "detected" test result who have pancreatic cancer diagnosed via imging in relation to all individuals in the intervention arm who had pancreatic cancer diagnosed.
Specificity of the Avantect test | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  The proportion of participants in the intervention arm with one or more Avantect "not detected" test results, and no Avantect "detected" results, who did not have a pancreatic cancer diagnosis in relation to all individuals in the intervention arm who did not have a pancreatic cancer diagnosis.
Resectability rate of pancreatic cancer | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  The proportion of pancreatic cancers deemed resectable by the study MDT divided by the number of pancreatic cancers and will be compared between arms.

SECONDARY OUTCOMES:
Stage shift | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  The proportion of pancreatic cancers cases diagnosed at stage I/II vs III/IV between the intervention and control arms. A proportion of 60% (44/73 PCs) is expected in the intervention arm versus 35% (26/73 PCs) in the control arm, which provides 90% power at a one-sided alpha of 0.05. Stage shift will be considered successful if the proportion in the intervention arm is higher than the rate in the control arm at a one-sided p-value of 0.05.
Positive Predictive Value (PPV) of Avantect test in detecting pancreatic cancer (PC) | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  Percentage of participants with an Avantect "detected" result who have pancreatic cancer diagnosed. The analysis will be conducted within the intervention arm. With a sample size of 7,500, PC prevalence of 1%, and 2.5% lost from the per protocol population, there will be an expected 410 individuals with an Avantect "detected - abnormal" result. 11.6% (48/410) are expected to have a PC. PPV will be considered successful if a null PPV of 5% can be ruled out at a one-sided p-value of 0.05.
Negative Predictive Value (NPV) of Avantect test in ruling out pancreatic cancer (PC) | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  Percentage of participants with no Avantect "detected" test result who have no diagnosis of pancreatic cancer. The analysis will be conducted within the intervention arm with a sample size of 7,500, PC prevalence of 1%, and 2.5% lost from the per protocol population, will be an expected 6,902 individuals without an Avantect "detected - abnormal" result. 99.6% (6,877/6,902) are expected to not have a diagnosis of PC. NPV will be considered successful if a null NPV of 99% can be ruled out at a one-sided p-value of 0.05.
Resection rate of pancreatic cancer | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  Percentage of participants with pancreatic cancer who underwent resection. The analysis will be conducted by comparing resection between the intervention and control arms. With a sample size of 15,000, PC prevalence of 1%, and 2.5% lost to follow-up, there will be an expected 73 cases of PC in each arm. It is assumed that 5% of those deemed resectable will not undergo resection, for an expected rate of 38% (28/73) in the Intervention arm versus 13% (9/73) in the control arm. Resection rate will be considered successful if the proportion in the intervention arm is higher than the rate in the control arm at a one-sided p-value of 0.05.

OTHER OUTCOMES:
Time-to-event outcomes | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  To estimate the time from new onset diabetes diagnosis to pancreatic cancer diagnosis. This will be analysed within intervention arm.
Overall survival | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  To estimate the overall survival of study participants. This will be compared between intervention and control arm.
Effect of the Avantect test on state anxiety over time | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  To assess the effect of the Avantect test on state anxiety over time. This will be compared between intervention and control arm.
High-grade neoplasia | Stage 1 analysis will be carried out 6 months after the T1 visit for 3,200 participants in the intervention arm. Stage 2 analysis will be carried out after 3-year follow-up data has been collected for all 15,000 participants.
  To investigate the performance characteristics for high-grade neoplasia. This will be analysed within intervention arm.

CONTACTS AND LOCATIONS:
Locations (14):
- United Kingdom (14):
  - Brockwood Medical Practice, Brockham, Surrey
  - Integrated Care Partnership/ The Old Cottage Hospital, Epsom, Surrey
  - Warlingham Green Medical Practice, Warlingham, Surrey
  - Bournemouth Research Hub, Bournemouth
  - Willesden Medical Centre, London
  - South Westminster Centre, London
  - The Cuckoo Lane Practice, London
  - King's Mill Hospital (Sherwood Forest) Research Van, Nottingham
  - Portsmouth Research Hub, Portsmouth
  - Pembroke Centre (Hillingdon), Ruislip
  - Southampton Research Hub (Shirley Research Hub), Southampton
  - Moorgreen Hospital, Southampton
  - Civic Centre, Uxbridge
  - Weymouth Research Hub, Weymouth

REFERENCES:
- See also: Related Info — https://safe-d.uk/